CLINICAL TRIAL: NCT04533048
Title: A Phase I Clinical Study to Evaluate the Safety, Tolerability, Pharmacokinetic Characteristics and Immunogenicity of a Single Dose of MW33 Injection in Healthy Subjects
Brief Title: A Clinical Study to Evaluate MW33 Injection
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Mabwell (Shanghai) Bioscience Co., Ltd. (Industry)
Collaborators: Shanghai Public Health Clinical Center (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MW33-2020-CP101
Record Dates: First submitted 2020-08-22; First posted 2020-08-31 (Actual); Last update posted 2021-02-26 (Actual); Status verified 2021-02

CONDITIONS: Covid19
MeSH Terms: conditions — COVID-19

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- MW33 (Experimental)
  Interventions: Combination Product: MW33 injection
- Placebo (Experimental)
  Interventions: Combination Product: MW33 injection placebo

INTERVENTIONS:
Combination Product: MW33 injection — a recombinant fully human antibody to coronavirus
  Arms: MW33
Combination Product: MW33 injection placebo — Placebo
  Arms: Placebo

SUMMARY:
This randomized, double-blind, placebo-controlled, single-dose escalation trial will be conducted to evaluate the safety, tolerability, immunogenicity, pharmacokinetic and pharmacodynamic characteristics of a single dose of MW33 injection at different doses given to healthy subjects to provide a basis for exploration of the therapeutic and preventive effects of MW33 against neocoronavirus in human.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects are fully aware of the purpose, nature, methods and possible adverse reactions of the study, voluntarily serve as subjects, and sign the informed consent form before the start of any study procedures, and ensure that he/she will participate in any procedures in the study in person;
2. Subjects are able to communicate well with the investigator and understand and comply with the requirements of the study;
3. The subject has no history of chronic or serious diseases involving the cardiovascular, liver, kidney, respiratory, blood and lymphatic, endocrine, immune, psychiatric, neurological, gastrointestinal system, and has a good general health condition;
4. Subjects (including male subjects) do not have a pregnancy plan, voluntarily take effective contraceptive measures during the screening period and the next 6 months, and have no sperm and egg donation plans, and shall voluntarily take non-pharmaceutical contraception measures during the trial period;
5. Male or female subjects aged 18 to 45 years (including 18 and 45 years);
6. Weight ≥ 50.0 kg for males, or weight ≥ 45.0 kg for females, and body mass index (BMI) in the range of 19.0 ~ 26.0 kg/m2 (including cut-off value);
7. Vital signs, physical examination, clinical laboratory tests (hematology, urinalysis, blood biochemistry, blood transfusion, coagulation function, pregnancy test [female], alcohol and drug screening, etc.), 12-lead electrocardiogram, chest X-ray and abdominal B-ultrasonography show no abnormalities or abnormalities without clinical significance.

Exclusion Criteria:

1. Health status: clinically significant histories of heart, liver, kidney, digestive tract, nervous system, respiratory system, blood and lymphatic system, immune system, mental, metabolic, and bone abnormalities.
2. Subjects who have a history of allergies to biological agents or any drug components; those who have a history of allergies and judged by the investigator to be ineligible for enrollment.
3. Those who have undergone surgery within 3 months prior to screening, or who plan to undergo surgery during the study, or who have undergone surgery that affects drug absorption, distribution, metabolism, and excretion.
4. Those who cannot tolerate venipuncture or have a history of needle-sickness and blood-sickness.
5. Those who have a history of drug abuse within 6 months prior to screening.
6. Use of illicit drugs within 3 months prior to screening.
7. Those who donated blood within 3 months prior to screening (including component blood), or massive blood loss (≥ 200 mL), or blood transfusions or use of blood products.
8. Subject (female) who is pregnant or lactating at screening or during the trial.
9. Subjects have a fertility plan or sperm or egg donation plan at screening and within the next 6 months.
10. Use of any prescription, over-the-counter, or Chinese herbal medicines within 2 weeks prior to screening.
11. Those who have been vaccinated within 4 weeks prior to screening or who are scheduled to be vaccinated during the study.
12. Those who have smoked more than 5 cigarettes per day within 3 months prior to screening, or who cannot stop using any tobacco products during the trial.
13. Those who have consumed more than 14 units of alcohol per week (1 unit of alcohol ≈ 360 mL of beer or 45 mL of spirits containing 40% alcohol or 150 mL of wine) within 3 months prior to screening, or who cannot abstain from alcohol during the trial.
14. Those who have special dietary requirements and cannot accept a standard diet.
15. Those who have participated in drug clinical trials and used investigational drugs within 3 months prior to screening.
16. Those who have previously used immunosuppressants or monoclonal antibodies for any reason.
17. Those with abnormal vital signs with clinical significance based on reference normal range (including cut-off values): sitting systolic blood pressure 90-139 mmHg, diastolic blood pressure 60-89 mmHg, pulse 60-100 beats/min, body temperature (ear temperature) 35.4-37.7 °C, respiration 16-20 breaths/min. The specific situation will be comprehensively determined by the investigator.
18. Those with abnormalities in laboratory tests and auxiliary examinations that are judged by the investigator to be clinically significant.
19. Those who have one or more clinically significant tests of hepatitis B virological markers, hepatitis C virus antibodies, anti-human immunodeficiency virus antibodies, or anti-Treponema pallidum-specific antibodies.
20. Female subjects with a positive urine or blood pregnancy test at screening.
21. Alcohol breath test results greater than 0.0 mg/100 ml or positive drug screening (morphine, icenarcotics [methamphetamine], ketamine, ecstasy [methylenedioxyamphetamine], cannabis [tetrahydrocannabinolate]).
22. Those who have acute illness from screening to day -1 admission.
23. Those who have taken any prescription, over-the-counter, Chinese herbal medicines from screening to day -1 admission.
24. Subjects who is inappropriate to participate in the trial due to any reasons as determined by the investigator.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2020-08-07 (Actual); Primary Completion 2020-11-16 (Actual); Study Completion 2020-12-02 (Actual)

PRIMARY OUTCOMES:
Adverse Event | 12 weeks
  safety evaluation
Serious Adverse Event | 12 weeks
  safety evaluation

CONTACTS AND LOCATIONS:
Locations (1):
- Shanghai Public Health Clinical Center, Shanghai, Shanghai Municipality, China

REFERENCES:
- [Derived] Kreuzberger N, Hirsch C, Chai KL, Tomlinson E, Khosravi Z, Popp M, Neidhardt M, Piechotta V, Salomon S, Valk SJ, Monsef I, Schmaderer C, Wood EM, So-Osman C, Roberts DJ, McQuilten Z, Estcourt LJ, Skoetz N. SARS-CoV-2-neutralising monoclonal antibodies for treatment of COVID-19. Cochrane Database Syst Rev. 2021 Sep 2;9(9):CD013825. doi: 10.1002/14651858.CD013825.pub2. PMID 34473343
- [Derived] Meng X, Wang P, Xiong Y, Wu Y, Lin X, Lu S, Li R, Zhao B, Liu J, Zeng S, Zeng L, Wu Y, Lu Y, Zhang J, Liu D, Wang S, Lu H. Safety, tolerability, pharmacokinetic characteristics, and immunogenicity of MW33: a Phase 1 clinical study of the SARS-CoV-2 RBD-targeting monoclonal antibody. Emerg Microbes Infect. 2021 Dec;10(1):1638-1648. doi: 10.1080/22221751.2021.1960900. PMID 34346827